CLINICAL TRIAL: NCT05717192
Title: Bronchoscopic Lung Volume Reduction in Severe Emphysema Using Thermoablation
Brief Title: BENTO - Bronchoscopic Lung Volume Reduction in Severe Emphysema Using Thermoablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDR-0002
Record Dates: First submitted 2022-12-19; First posted 2023-02-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-12

CONDITIONS: Emphysema or Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- InterVapor®-System (Active Comparator): The intervention to be tested is bronchoscopic lung volume reduction (BTVA) using thermal ablation (InterVapor®, Uptake Medical, California, USA). This is performed in addition to standard conservative therapy in accordance with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines. The intervention can consist of a maximum of two partial interventions
  Interventions: Device: InterVapor®-System
- Standard of care (No Intervention): Standard conservative therapy in accordance with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines without the use of a BTVA (patient-specific documentation of therapeutic measures).

INTERVENTIONS:
Device: InterVapor®-System — The InterVapor System uses heated water vapor to ablate the airways and parenchyma within targeted regions of the lung. Lung remodeling occurs after an initial localized inflammatory response and a subsequent healing and repair. The remodeling of the tissue results in reductions in tissue and air volume in the targeted regions of the lung. The remodeled lung tissue does not re-inflate as a result of collateral ventilation.
  The lung volume reduction of diseased hyper-inflated lung segments after InterVapor treatment is expected to increase elastic recoil by reducing the most compliant segments of the lung, decompressing segments of healthier lung allowing for alveolar recruitment, and improving the mechanical efficiency of the respiratory muscles. These mechanical changes are anticipated to improve pulmonary function, exercise capacity and quality of life.
  Arms: InterVapor®-System

SUMMARY:
Prospective, 2-arm, randomised (2:1), multicentre, open-label clinical trial in patients with severe emphysema. The intervention arm will be treated with Bronchoscopic lung volume reduction in severe emphysema using thermoablation.The interventional treatment (bronchoscopic lung volume reduction) is compared with the usual conservative standard therapy (GOLD guidelines).

DETAILED DESCRIPTION:
Currently, there is less data on the use of bronchoscopic thermoablation (BTVA) for the treatment of patients with emphysema. However, the current studies suggest with a high degree of certainty that bronchoscopic lung volume reduction for severe emphysema using thermoablation has the potential to be a necessary treatment alternative. The trial study should therefore contribute to proving the benefit of this procedure as an effective and safe treatment option in order to guarantee emphysema patients sufficient, appropriate and economical care, taking into account evidence-based medical knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 40 years and ≤ 75 years
* Written informed consent obtained from the patient
* Severe emphysema with indication for BTVA:
* bilateral heterogeneous emphysema of the upper lobes in GOLD stage 3/4 and
* evidence of severe emphysema in high-resolution computed tomography (not older than 6 months prior to inclusion) and
* functional evidence of severe pulmonary hyperinflation and
* FEV1 post lysis between 20% and < 45% (calculated) and
* Total lung capacity (TLC) ≥ 100% (calculated) and
* Residual volume (RV) > 175% (calculated) and
* arterial blood gas values of: PaCO2 ≤ 50 mmHg; PaO2 > 50 mmHg on room air and
* marked dyspnoea with a score ≥ 2 on the Medical Research Council modified scale (mMRC) and
* 6-minute walk test > 140 metres
* Patient-specific, pre-interventional exhaustion of conservative treatment options
* optimised medical therapy (according to the GOLD guidelines) and
* Non-smoker for 6 months prior to inclusion
* Evidence of completed pulmonary and geriatric rehabilitation in the last 4 years
* ≥ 6 weeks outpatient or
* ≥ 3 weeks inpatient or
* Individual Participation in regular physical activities that go beyond the activities of daily living (e.g. a walking programme)
* According to the investigator's assessment mentally and physically able to participate in the study procedures and visits
* Indication within the framework of an interdisciplinary case conference with specialists in pneumology, radiology and thoracic surgery in accordance with §3 of the guideline on quality assurance measures in accordance with § 136 Paragraph 1 Sentence 1 Number 2 SGB V for inpatient care with bronchoscopic lung volume reduction procedures for severe emphysema (QS-RL BLVR).

Exclusion Criteria:

* Any condition that would interfere with the conduct of the clinical trial follow-up or bronchoscopy or affect the outcome of the clinical trial
* DLCO < 20% (calculated)
* Body mass index (BMI) < 18 kg/m2 or > 32 kg/m2
* Pulmonary hypertension
* Peak systolic PAP > 45 mmHg or mean PAP > 25 mmHg
* Right heart catheter measurements are considered authoritative over echocardiogram measurements
* Clinically significant bronchiectasis
* Pneumothorax or pleural effusions within the last 6 months
* Heart and/or lung transplantation, surgical lung volume reduction (LVRS), bullectomy, lobectomy or pneumonectomy, pleurodesis or any surgery in the target lobes (upper lobes).
* Recent respiratory infection or COPD exacerbation in the last 6 weeks
* Unstable COPD (any of the following conditions):
* >3 COPD-related hospitalisations requiring antibiotics in the last 12 months
* COPD-related hospital stay in the last 3 months
* daily use of systemic steroids, > 5 mg prednisolone
* Single large bulla (defined as > 1/3 of the volume of the lobe) in the upper lobe or paraseptal emphysema distribution in the lobe being treated
* Coagulopathy or current use of anticoagulants
* Patients with current endobronchial valves or with valves explanted less than 6 months ago in the target lobe in a segment to be treated with InterVapor®.
* Patients with implanted, endobronchial coils (coils)
* Patients with previous endobronchial polymer/adhesive treatment
* Patients with immune system disorders or concomitant diseases that necessitate the use of immunosuppressants of clinical relevance
* History of any of the following conditions:
* Myocardial infarction or acute coronary syndrome in the previous year
* Hospitalisation for left heart failure in the last year
* clinically leading asthma disease or alpha-1-antitrypsin deficiency
* Known sensitivity to medications required to perform bronchoscopy
* Life expectancy < 12 months
* Newly prescribed morphine derivatives within the last 4 weeks
* Pregnancy at the time of inclusion

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported disease-specific quality of life | 9 months
  Change in patient-reported, disease-specific quality of life based on St. George's Respiratory Questionnaire (SGRQ-C) between randomisation and 9-month visit.
  The instrument has 3 domains (activity, symptoms, and impacts) and a total score. A Total and three-component scores are calculated: Symptoms; Activity; Impacts. Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100. Each component of the questionnaire is scored separately. Sum of maximum possible weights for each component and Total: Symptoms 566.2, Activity 982.9, Impacts 1652.8. Total (sum of maximum for all three components) 3201.9 Higher weights indicate worse outcomes. The difference in the domain scores and total score at follow-up visits relative to baseline will be calculated and reported.

SECONDARY OUTCOMES:
Vital status | 3, 9 and 12 months
  alive/dead
Change in FEV 1 | 3, 9 and 12 months
  Change in forced expiratory pressure (FEV 1) in litres and percent
Change in RV | 3, 9 and 12 months
  Change in residual volume in litre and percent.
Change in patient-reported, disease-specific quality of life | 3, 9 and 12 months
  Change in patient-reported, disease-specific quality of life based on St. George's Respiratory Questionnaire (SGRQ-C) between randomisation and 9-month visit.
  The instrument has 3 domains (activity, symptoms, and impacts) and a total score. A Total and three-component scores are calculated: Symptoms; Activity; Impacts. Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100. Each component of the questionnaire is scored separately. Sum of maximum possible weights for each component and Total: Symptoms 566.2, Activity 982.9, Impacts 1652.8. Total (sum of maximum for all three components) 3201.9 Higher weights indicate worse outcomes. The difference in the domain scores and total score at follow-up visits relative to baseline will be calculated and reported.
Serious Adverse Events | 3, 9 and 12 months
  Rate of serious adverse events
6-minute walk test (6MWT) | 3, 9 and 12 months
  Measures the distance (meter) in a 6-minute walk test.
Severe excacerbations | 3, 9 and 12 months
  Rate of severe exacerbations
Mortality | 3, 9 and 12 months
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Charité Campus Benjamin Franklin, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe gGmbH Klinik für Anthroposophische Medizin, Berlin
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik II, Bonn
  - Pneumologische Universitätsklinik Ruhrlandklinik, Essen
  - Universitätsklinikum Halle (Saale), Halle
  - Thoraxklinik University of Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Asklepios Klinik Langen, Klinik für Innere Medizin III, Langen
  - KlinKlinikuim Lüdenscheid, Klinik für Pneumologie, internistische Intensivmedizin, Infektiologie und Schlafmedizin, Lüdenscheid
  - Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Helios Hanseklinikum Stralsund, Stralsund

IPD SHARING:
Plan to Share IPD: No
Data Sharing Processes
  All subject-level clinical, laboratory, and quality of life data will be preserved and shared with the Sponsor via eCRF. Shared data will be deidentified and original data will be main-tained at the investigator's site. Study design, recruitment progress and final results will be documented at clinicaltrials.gov. The trial data will be passed on to the extent permitted by the patient´s informed consent. Upon completion of the study, individual participant data will not be made available on data sharing repositories.
  The steering committee will decide on sharing study data upon reasonable request.

REFERENCES:
- [Derived] Kontogianni K, Darwiche K, Huebner RH, Hassinger F, Riemer T, Herth FJ, Brock J. Design of the multicentre randomised controlled BENTO trial to demonstrate patient-relevant benefit of bronchoscopic lung volume reduction using thermal vapour ablation in the German healthcare system for patients with upper lobe emphysema: a study protocol. BMJ Open. 2024 May 28;14(5):e080518. doi: 10.1136/bmjopen-2023-080518. PMID 38806430